CLINICAL TRIAL: NCT03427554
Title: A Multi-center, Double-Blind, Randomized, Placebo Controlled, Parallel-Group Study, Comparing TRETINOIN CREAM, 0.1% to RETIN-A® (TRETINOIN) CREAM, 0.1% and Both Active Treatments to a Placebo Control in the Treatment of Acne Vulgaris
Brief Title: To Evaluate the Therapeutic Equivalence and Safety of TRETINOIN CREAM, 0.1% and RLD in the Treatment of Acne Vulgaris
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Sun Pharmaceutical Industries, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TRTC 1622
Record Dates: First submitted 2018-01-29; First posted 2018-02-09 (Actual); Last update posted 2018-05-18 (Actual); Status verified 2018-05

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — Tretinoin

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Tretinoin cream 0.1% (Experimental): Once daily at home, to apply the entire affected areas of the face.
  Interventions: Drug: Tretinoin cream 0.1%
- RETIN-A® Cream (Active Comparator): Once daily at home, to apply the entire affected areas of the face.
  Interventions: Drug: RETIN-A® Cream
- Vehicle of the test product (Placebo Comparator): Once daily at home, to apply the entire affected areas of the face.
  Interventions: Drug: Vehicle of the test product

INTERVENTIONS:
Drug: Tretinoin cream 0.1% — Tretinoin cream 0.1% (Taro Pharmaceuticals Inc.)
  Other Names: Tretinoin
  Arms: Tretinoin cream 0.1%
Drug: RETIN-A® Cream — RETIN-A® (Tretinoin) Cream (Valeant)
  Other Names: Tretinoin
  Arms: RETIN-A® Cream
Drug: Vehicle of the test product — Vehicle for Tretinoin cream 0.1% (Taro Pharmaceuticals Inc.)
  Other Names: Placebo
  Arms: Vehicle of the test product

SUMMARY:
Bioequivalence study comparing Tretinoin Cream, 0.1% to RETIN-A®.

DETAILED DESCRIPTION:
A Multi-center, Double-Blind, Randomized, Placebo controlled, Parallel-Group study, comparing TRETINOIN CREAM, 0.1% (TARO PHARMACEUTICALS U.S.A., INC.) to RETIN-A® (TRETINOIN) CREAM, 0.1% (VALEANT) and both active treatments to a Placebo Control in the treatment of Acne Vulgaris

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or non pregnant female aged ≥ 12 and ≤ 40 years with a clinical diagnosis of acne vulgaris.
* Subjects must have a definite clinical diagnosis of acne vulgaris severity grade 2, 3, or 4 as per the Investigator's Global Assessment (IGA).
* Subjects must be willing and able to understand and comply with the requirements of the protocol, including attendance at the required study visits.

Exclusion Criteria:

* Female Subjects who are pregnant, nursing or planning to become pregnant during study participation.

Ages: 12 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 455 (Actual)
Dates: Start 2017-08-21 (Actual); Primary Completion 2018-01-26 (Actual); Study Completion 2018-01-26 (Actual)

PRIMARY OUTCOMES:
Demonstration of Bioequivalence | 12 weeks
  Demonstration of Bioequivalence in Percent change in inflammatory and non-inflammatory lesion counts

CONTACTS AND LOCATIONS:
Overall Officials: Zaidoon A Al-Zubaidy, Study Director — Catawba Research
Locations (1):
- Catawba Research, LLC, Charlotte, North Carolina, United States